CLINICAL TRIAL: NCT01562132
Title: An Open Label Randomized Controlled Phase IIb Trial to Determine the Safety of Oral Fluconazole in Combination With Flucytosine as Compared to Fluconazole Alone
Brief Title: Safety Study of Fluconazole in Combination With Flucytosine for the Treatment of Early Cryptococcal Infection
Acronym: SToP-Crypto
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped in accordance with pre-specified stopping rules for poor recruitment.
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Kenya Medical Research Institute (Other); Bausch Health Americas, Inc. (Industry); University of Nairobi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1307012426; R21NS077858-01 (NIH)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cryptococcal Infection Disseminated
Keywords: cryptococcus; HIV
MeSH Terms: interventions — Flucytosine; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5FC plus fluconazole (Experimental): Combination therapy with oral fluconazole and flucytosine
  Interventions: Drug: Flucytosine and fluconazole
- fluconazole alone (Active Comparator): Fluconazole monotherapy
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Flucytosine and fluconazole — Flucytosine 100mg/kg/day in 4 divided doses orally for 14 days given in combination with fluconazole 1200mg orally once daily for 14 days, followed by 800mg orally once daily for 8 weeks, followed by 200mg orally once daily
  Other Names: Ancobon; Diflucan
  Arms: 5FC plus fluconazole
Drug: Fluconazole — fluconazole 1200mg orally once daily for 14 days, followed by 800mg orally once daily for 8 weeks, followed by 200mg orally once daily
  Other Names: Diflucan
  Arms: fluconazole alone

SUMMARY:
The purpose of this study is to determine if treatment with two medicines in combination (fluconazole and flucytosine) is safe as compared with one medicine alone (fluconazole) for the treatment of an early infection with a fungus called cryptococcus.

DETAILED DESCRIPTION:
Currently there is wide variation in practice and little evidence to guide the treatment of early cryptococcal infection in HIV-infected individuals with advanced immunosuppression. However, epidemiologic studies suggest that this may be a promising novel approach to decrease the mortality due to cryptococcal meningitis (CM), the second leading cause of death among HIV-infected individuals in many resource-limited settings. Screening asymptomatic HIV-infected individuals with advanced immunosuppression for serum cryptococcal antigen (CrAg) clearly identifies a population at high risk of CM and death and is a feasible screening method for resource-limited settings. However, screening with serum CrAg alone without additional diagnostic studies identifies a heterogeneous clinical population with early cryptococcal infection, many of whom already have sub-clinical meningeal infection or fungemia. The mainstay of anti-cryptococcal therapy in resource-limited settings is oral fluconazole though preliminary evidence suggests this is not an effective treatment. Thus, there is a critical need for potent therapies that (1) can be safely administered in resource-limited settings and (2) are effective in a heterogeneous population of HIV-infected individuals with advanced immunosuppression and early cryptococcal infection who are initiating anti-retroviral therapy (ART).

This single center, open-label, randomized Phase IIb study is being conducted to assess the safety and estimate the efficacy of oral fluconazole in combination with flucytosine for the treatment of early cryptococcal infection. The study will be based at two sites supported by Family AIDS Care and Education Services (FACES) in Western Kenya. A consecutive sample of 100 HIV-infected adults with CD4 cell count ≤100 cells/µl and serum CrAg titer ≥1:2 who have no signs or symptoms of severe, systemic cryptococcal infection will be enrolled. At enrollment, specimens from participants will be cultured for evidence of Cryptococcus neoformans. Individuals who meet inclusion and exclusion criteria and consent to participate in the study will be randomized to combination therapy with oral fluconazole (1200mg/day) plus flucytosine (100mg/kg/day) or fluconazole alone for the fourteen days of therapy. Subsequently both groups will receive anti-retroviral therapy as well as fluconazole 800mg/day for 8 weeks followed by 200mg/day. The primary safety endpoint will be the incidence of treatment-related adverse events and serious adverse events. The primary efficacy endpoint will be survival at 12 weeks.

In addition, we will offer additional diagnostic testing and aim for 50% participation, approximately 25 individuals from each arm. We will perform a battery of diagnostic tests including chest radiography, fungal cultures in blood, sputum, urine, stool and cerebrospinal fluid (CSF), cryptococcal antigen testing in the CSF, and gram stain, Ziehls-Nielsen stain and India Ink staining of CSF sediment. Anti-fungal susceptibility testing via broth microdilution and polymerase chain reaction serotyping and mating type analysis will be performed on clinical isolates.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* Age > 18 years
* HIV infection as confirmed by HIV-antibody test as per Kenyan guidelines
* CD4+ T-cell count ≤100 cells/µl
* Serum CrAg titer≥1:2
* Able to travel to district hubs (Sindo District Hospital, Lumumba Health Centre) for regular study visits

Exclusion Criteria:

* clinical meningitis:
* clinical sepsis:
* hemiparesis, aphasia, visual field deficit or other finding on neurological examination localizable to the central nervous system
* a history of culture proven or suspected (cryptococcal antigen present) cryptococcal meningitis
* a history of stroke or other infection of the central nervous system
* a seizure within the last 2 months
* currently taking or ever taken antiretroviral therapy
* currently taking anti-tuberculous therapy
* currently or recently (<2 months) prescribed fluconazole, itraconazole, clotrimazole troches, amphotericin or other oral anti-fungal medications
* pregnant or breast-feeding
* alanine aminotransferase concentration more than 3 times the upper limit of normal
* neutrophil count <1000x103 cells/mL
* hemoglobin <8g/dL
* platelet count <100,000x 103 platelets/mL
* creatinine clearance ≤50 ml/min
* individuals with active heavy alcohol use or active recreational drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Claire L Meyer, MD, MSHS, Principal Investigator — University of California, San Francisco; Mark A Jacobson, MD, Principal Investigator — University of California, San Francisco; Judith K Kwasa, MBChB MMed, Principal Investigator — University of Nairobi
Locations (2):
- Kenya (2):
  - Family AIDS Care and Education Services, Kisumu, Nyanza
  - Family AIDS Care and Education Services, Sindo, Nyanza

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5FC Plus Fluconazole | Fluconazole Alone
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5FC Plus Fluconazole | Fluconazole Alone | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 36 [28 to 49] | 31 [26 to 58] | 33.5 [26 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Kenya | 3 | 3 | 6
CD4+ T-cell Count [Median (Full Range); unit: cells/microliter] | 22 [18 to 56] | 13 [3 to 16] | 17 [3 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Alive at 12 Weeks
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | 5FC Plus Fluconazole | Fluconazole Alone
Number analyzed (Participants) | 3 | 3
participants | 2 | 2

2. Secondary Outcome: Number of Participants Alive at 2 Weeks
Time Frame: 2 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Survival at 24 Weeks
Time Frame: 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Number of Individuals Who Develop Cryptococcal Meningitis
Description: Clinical meningitis AND at least one of the following: cryptococcal antigen in the cerebrospinal fluid (CSF), cryptococcal organisms on India Ink stain, or fungal culture of CSF.
  Clinical meningitis will be defined as:
  * fever>39.0°C, AND
  * severe headache, AND
  At least one of the following:
  * meningismus,
  * photophobia,
  * new onset seizure,
  * focal neurological deficit localizable to the central nervous system
  * papilledema
  * confusion, delirium, or decreased level of consciousness.
Time Frame: 24 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Number of Individuals Who Develop Immune Reconstitution Inflammatory Syndrome Due to Cryptococcus
Description: Individuals who develop clinical meningitis without evidence of fungal, bacterial, or parasitic (e.g. malaria) organisms in the cerebrospinal fluid. Clinical meningitis will be defined as:
  * fever>39.0°C, AND
  * severe headache, AND
  * At least one of the following:
  * meningismus,
  * photophobia,
  * new onset seizure,
  * focal neurological deficit localizable to the central nervous system
  * papilledema
  * confusion, delirium, or decreased level of consciousness.
Time Frame: 24 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Achieve Targeted Recruitment, Retention and Adherence Rates
Time Frame: 24 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Proportion of Individuals Requiring Treatment Discontinuation
Time Frame: 4 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Proportion of Individuals Requiring Dose Reduction
Time Frame: 24 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Number of Individuals With Treatment Related Adverse Events
Time Frame: 24 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Number of Individuals With Treatment Related Serious Adverse Events
Time Frame: 24 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Cryptococcal Meningitis-free Survival at 24 Weeks
Description: as for outcome 4
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 5FC Plus Fluconazole | Fluconazole Alone
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5FC Plus Fluconazole (N=3) | Fluconazole Alone (N=3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) — Grade 1
Unintentional Weight Loss (General disorders) | 1 (1) | 0 (0) — Grade 2
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less